CLINICAL TRIAL: NCT05148351
Title: Validity of an iPhone App to Detect Frailty and Sarcopenia Syndromes in Community Dwelling Older Adults: Protocol for a Diagnostic Accuracy Study
Brief Title: Validity of an App to Detect Frailty and Sarcopenia Syndromes in Elderly
Status: Completed | Type: Observational
Sponsor: Catholic University of Murcia (Other)
Responsible Party: Principal Investigator, Alessio Montemurro, Principal Investigator, Catholic University of Murcia
Other Study IDs: Universidad Católica de Murcia
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Sarcopenia; Frailty Syndrome; Aging; Aged; Diagnosis
Keywords: Functional Capacity; Sit-to-Stand Test; Muscle Power; Chair rise
MeSH Terms: conditions — Sarcopenia; Frailty; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty and sarcopenia are two age-related syndromes which can result in adverse health-related events. The combination of both is more predictive of mortality than either condition alone. These conditions can be reversed through an early detection and appropriate interventions. Nevertheless, scientific community highlights the lack of cheap, portable, rapid and easy-to-use tools for detecting frailty and sarcopenia in combination. The aim of this study is to validate an iPhone App to detect frailty and sarcopenia syndromes in community dwelling older adults. This is a protocol study of a retrospective diagnostic test accuracy study which will include at least 400 participants older than 60 years recruited from elderly social centers of Murcia city. Researchers will recollect data of health status, dependency, cognitive status, and functional capacity of the participants. The index test will consist in the measurement of muscle power exerted during a single Sit-to-stand through an App (iPhone), combined with calf and mid-upper arm circumference. The reference standard will be frailty syndrome and sarcopenia assessed according to Fried's phenotype and to the European Working Group on Sarcopenia in Older People 2 (EWGSOP2) (2019) recommendations, respectively. Sensitivity, specificity, positive predictive value, negative predictive values, and area under the curve will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults living in the Region of Murcia

Exclusion Criteria:

* Barthel Index < 90 pts.
* Mini-Cog test < 3 pts.
* Severe cardiovascular problems
* Pacemaker
* Automatic defibrillator

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 400 community-dwelling older adults, older than 60 y/o and living in the Region of Murcia (Spain) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Muscular power | Cross-sectional baseline
  Muscular power generated by participants will be measured using an App (Sit-to-stand App version 1.1) installed on an iPhone (Apple Inc., USA).
  During the execution, subjects will sit on a rigid chair with their arms crossed over their chest with the hip, knee and ankle joints at approximately 90 degrees. Subjects will be asked to stand-up as fast as possible. Participants will complete three STS repetitions. No footwear will be allowed during the test.
Frailty Syndrome | Cross-sectional baseline
  Frailty Syndrome will be assessed according to Fried's Phenotype, which focuses on:
  1. Handgrip strength
  2. Usual gait speed
  3. Weight loss
  4. Exhaustion
  5. Physical activity levels
  Subjects who will result positive to three out of five criteria will be considered as "frail", whereas if they will result positive to only one or two of them they will be considered as "pre-frail". The absence of each criteria will be necessary to define a subject as "robust".
Sarcopenia | Cross-sectional baseline
  Sarcopenia will be assessed according to the recommendation provided by the European Working Group on Sarcopenia in Older People 2 (EWGSOP2) (2019). This guideline focuses on the assessment of:
  1. Leg muscle strength
  2. Muscle mass quantity
  3. Physical performance
  The presence of low muscle strength levels will be considered as "probable sarcopenia"; the presence of low muscle mass and strength levels will be considered as "confirmed sarcopenia"; finally, the presence of the three criteria will be considered as "severe sarcopenia".
Calf and mid-upper arm circumference | Cross-sectional baseline
  Researchers will measure subjects' calf and mid-upper arm circumference using a tape measure.

SECONDARY OUTCOMES:
Subjects' clinical status | Cross-sectional baseline
  Subjects' clinical status will be assessed through a list of questions regarding:
  * socioeconomic level
  * educational level
  * chronic pathologies
  * smoking habits
  * polypharmacy
  * depression
  * number of falls
  * hospitalization
  * self-perceived health status

CONTACTS AND LOCATIONS:
Overall Officials: Juan D Ruiz-Cárdenas, Study Director — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruiz-Cardenas JD, Rodriguez-Juan JJ, Martinez-Garcia MDM, Montemurro A. Comparing Sarcopenia Definitions and Muscle Power Reduction: Associations with Health Outcomes in Spanish Community-Dwelling Older Adults. J Clin Med. 2024 Aug 23;13(17):4988. doi: 10.3390/jcm13174988. PMID 39274199
- [Derived] Ruiz-Cardenas JD, Montemurro A, Martinez-Garcia MDM, Rodriguez-Juan JJ. Sit-to-Stand Video Analysis-Based App for Diagnosing Sarcopenia and Its Relationship With Health-Related Risk Factors and Frailty in Community-Dwelling Older Adults: Diagnostic Accuracy Study. J Med Internet Res. 2023 Dec 8;25:e47873. doi: 10.2196/47873. PMID 38064268
- [Derived] Montemurro A, Ruiz-Cardenas JD, Martinez-Garcia MDM, Rodriguez-Juan JJ. Validity of an iPhone App to Detect Prefrailty and Sarcopenia Syndromes in Community-Dwelling Older Adults: The Protocol for a Diagnostic Accuracy Study. Sensors (Basel). 2022 Aug 11;22(16):6010. doi: 10.3390/s22166010. PMID 36015771